CLINICAL TRIAL: NCT05524636
Title: Effects of Abdominal Wall Muscle Training With or Without Additional Peripheral Magnetic Stimulation on Subcutaneous Fat, Muscle Strength and Postural Control
Brief Title: Effects of Peripheral Magnetic Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Collaborators: Fotona d.o.o. (Industry)
Responsible Party: Principal Investigator, Nejc Sarabon, Professor, PhD, University of Primorska
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fotona
Record Dates: First submitted 2022-08-25; First posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Healthy
Keywords: subcutaneous fat, magnetic stimulation, abdominal muscles
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Experimental and control group
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Exercise with peripheral magnetic stimulation of the abdominal wall muscles
  Interventions: Device: Exercise with peripheral magnetic stimulation of the abdominal wall muscles
- Control (Active Comparator): Exercise without peripheral magnetic stimulation of the abdominal wall muscles
  Interventions: Other: Exercise of the abdominal wall muscles

INTERVENTIONS:
Device: Exercise with peripheral magnetic stimulation of the abdominal wall muscles — 8-week exercise program with peripheral magnetic stimulation, focused on abdominal wall muscles aiming to reduce subcutaneous fat, increase abdominal wall muscle strength and improve sitting postural control.
  Arms: Experimental
Other: Exercise of the abdominal wall muscles — 8-week exercise program focused on abdominal wall muscles aiming to reduce subcutaneous fat, increase abdominal wall muscle strength and improve sitting postural control.
  Arms: Control

SUMMARY:
Interventional study of the effectiveness of peripheral magnetic stimulation of the abdominal wall muscles in healthy individuals.

DETAILED DESCRIPTION:
Interventional 8-week study of the effectiveness of peripheral magnetic stimulation of the abdominal wall muscles in healthy individuals. The study will include an experimental and a control group.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults
* BMI between 25,0 and 29,9 kg/m2
* stable body mass with maximal variation of body mass of 2.2 kg a month prior to the inclusion in the study
* waist circumference above 80 cm for females and above 90 cm for males

Exclusion Criteria:

* invasive fat reduction procedures (e.g., liposuction and mesotherapy)
* weight loss supplements in the month prior to the participation in the study
* metal implant
* active implanted electrical device such as a cardiac pacemaker, cochlear implant, intrathecal pump, hearing aids, defibrillator, or drug delivery system

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Change in subcutaneous fat | Baseline, 4 weeks, 8 weeks, 12 weeks after baseline measurement
  Subcutaneous fat thickness in the abdominal area measured via ultrasound
Change in maximum isometric peak torque | Baseline, 4 weeks, 8 weeks, 12 weeks after baseline measurement
  Maximal voluntary isometric contraction of the abdominal muscles. The measurement will be normalized to the body weight (Nm/kg).
Change in sitting postural control | Baseline, 4 weeks, 8 weeks, 12 weeks after baseline measurement
  Sitting on an unstable surface for 30 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Nejc Šarabon, PhD, Principal Investigator — Fakulteta za vede o zdravju
Locations (1):
- University of Primorska, Izola, Primorska, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
Coded individual data will be uploaded on public scientific data repository.
Supporting Information: Study Protocol